CLINICAL TRIAL: NCT07054931
Title: AbVax: Combination Vaccination and Broadly Neutralising Antibody Therapy in HIV to Induce a Protective T-cell 'Vaccinal Effect' - a Randomised Phase II Clinical Trial
Brief Title: Combination Vaccination and Broadly Neutralising Antibody Therapy in HIV
Acronym: AbVax
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbVax; MR/Y008847/1 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2025-05-16; First posted 2025-07-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: HIV
Keywords: vaccination; broadly neutralising antibodies; HIV treatment

STUDY DESIGN:
Intervention Model Description: Participants are randomised to one of three arms. Participants in Arm A undergo a period of treatment interruption induced viraemia, followed by two bNAB infusions (GS-5423 and GS-2872). Participants in Arm B receive three HIV vaccines (one prime dose of two vaccines, ChAdOx1.tHIVconsv1 and ChAdOx2.HIVconsv62 and two booster doses of MVA.tHIVconsv4 after 4 and 16 weeks), followed by two bNAb infusions (GS-5423 and GS-2872). Participants in Arm C undergo a period of treatment interruption induced viraemia, followed by three HIV vaccines (one prime dose of two vaccines, ChAdOx1.tHIVconsv1 and ChAdOx2.HIVconsv62 and two booster doses of MVA.tHIVconsv4 after 4 and 16 weeks), followed by two bNAb infusions (GS-5423 and GS-2872). All participants then undergo a period of analytical treatment interruption where there responses to the interventions are measured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Participants in Arm A will undergo a period of treatment interruption induced viraemia followed by two infusions of broadly neutralising antibodies (GS-5423 and GS-2872). They will then stop ART for an analytical treatment interruption period to determine the clinical impact and to measure how long before any HIV virus returns to the blood.
  Interventions: Biological: GS-5423; Biological: GS-2872; Other: Treatment interruption induced viraemia
- Arm B (Active Comparator): Participants in Arm B will receive a combination of three HIV vaccines (one prime dose (ChAdOx1.tHIVconsv1 and ChAdOx1.HIVconsv62) followed by two booster doses of MVA.tHIVconsv4 at 4 weeks and 16 weeks), followed by two infusions of broadly neutralising antibodies, GS-5423 and GS-2872. They will then stop ART for an analytical treatment interruption period to determine the clinical impact and to measure how long before any HIV virus returns to the blood.
  Interventions: Biological: ChAdOx1.tHIVconsv1; Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv4; Biological: GS-5423; Biological: GS-2872
- Arm C (Active Comparator): Participants in Arm C will undergo a period of treatment interruption induced viraemia followed by a combination of three HIV vaccines (one prime dose (ChAdOx1.tHIVconsv1 and ChAdOx1.HIVconsv62) followed by two booster doses of MVA.tHIVconsv4 at 4 weeks and 16 weeks), followed by two infusions of broadly neutralising antibodies, GS-5423 and GS-2872. They will then stop ART for an analytical treatment interruption period to determine the clinical impact and to measure how long before any HIV virus returns to the blood.
  Interventions: Biological: ChAdOx1.tHIVconsv1; Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv4; Biological: GS-5423; Biological: GS-2872; Other: Treatment interruption induced viraemia

INTERVENTIONS:
Biological: ChAdOx1.tHIVconsv1 — solution for injection one dose of 2.5 x 10^10 vp/ml Arm B and Arm C
  Arms: Arm B; Arm C
Biological: ChAdOx1.HIVconsv62 — solution for injection one dose of 2.5 x 10^10 vp/ml Arm B and Arm C
  Arms: Arm B; Arm C
Biological: MVA.tHIVconsv4 — suspension for injection two doses of 1 x 10^8 vpu/ml Arm B and Arm C
  Arms: Arm B; Arm C
Biological: GS-5423 — Solution for infusion 2550 mg Arm A, Arm B and Arm C
Biological: GS-2872 — Solution for infusion 850 mg Arm A, Arm B and Arm C
Other: Treatment interruption induced viraemia — Participants pause ART before receiving vaccines and/or bNAbs Arm A and Arm C
  Arms: Arm A; Arm C

SUMMARY:
There is no cure for HIV infection. Antiretroviral therapy (ART) is widely available but requires daily, life-long intake. This can cause issues around side-effects, resistance, adherence and stigma. A new therapy, broadly neutralising antibodies, (bNAbs), may work as well as ART and may last longer - one dose can last six months. bNAbs appear to first target HIV viruses, then drive a protective immune response conferring long-term control, called the vaccinal effect. AbVax is a clinical trial to understand this effect and how to enhance it to give the strongest possible long-term protection for people living with HIV (PWH). The investigators are studying whether a combination of vaccines that attack HIV, a short period of treatment interruption induced viraemia (TIIV - stopping ART for a few weeks to allow a small amount of virus to return to the bloodstream) and bNABs will produce the most sustained immune protection.

DETAILED DESCRIPTION:
AbVax will recruit 48 otherwise healthy PWH aged 18-64. Participants will be randomised across three groups (arms) to determine the best combination of treatment. In Arm A, participants will undergo a period of TIIV, then receive two bNAb infusions. In Arm B, participants receive a combination of three HIV vaccines (one prime dose followed by two booster doses after 4 and 16 weeks), then are given two bNAb infusions. In Arm C, participants will undergo a period of TIIV, then receive the same vaccination combinations as Arm B, then receive two bNAb infusions. All participants then stop ART for an analytical treatment interruption (ATI) to determine the clinical impact and measure how long before any HIV returns to the blood. This allows the investigators to see if vaccines and TIIV add to the protection provided by bNAbs and by how much.

ELIGIBILITY:
Inclusion Criteria:

* PWH aged ≥18 to ≤64 years old at screening

  * Able to give informed written consent including consent to long-term follow-up
  * Willing and able to comply with visit schedule and provide blood sampling
  * Willing to consent to their HIV care team being informed of their participation and sharing relevant clinical information
  * Stable on oral ART with suppressed undetectable HIV pVL 'target not detected' (TND) using local assays for ≥ 1 years (a single viral load measurement >50 but <500 copies/ml during this time period is allowable)
  * No evidence of viral insensitivity to GS-2872 based on proviral sequencing
  * No significant co-morbidities according to the investigator's opinion
  * Nadir CD4 >200 cells/µl unless treatment commenced during documented acute seroconversion
  * Current CD4 count >500 cells/µl or CD4:CD8 ratio >1.0
  * On integrase inhibitor (INSTI) or boosted protease inhibitor (bPI) based regimen at time of randomisation. If previously on non-nucleoside reverse transcriptase inhibitor (NNRTI) must have switched at least 4 weeks prior to randomisation
  * Adequate haemoglobin (Hb ≥12 g/dL for males, ≥11 g/dL for females)
  * Weight ≥ 50kg
  * Has received at least 3 doses of vaccination against coronavirus (COVID-19), at least 4 weeks prior to randomisation
  * Has received current seasonal vaccination against Influenza*
  * People of childbearing potential** must agree to use hormonal contraception, intrauterine device, intrauterine hormone-releasing system, or otherwise practice complete abstinence*** from at least two weeks before the first Investigational Medicinal Product (IMP) administration, for at least 20 months after the last IMP administration, and until undetectable viral load on ART
  * All participants must agree to take precautions to prevent onward transmission of HIV (such as condoms or PrEP) whilst they are off ART and/or have a detectable viral load * Applicable during Influenza season (September-April inclusive). **Individuals capable of becoming pregnant are defined as those who are fertile, with childbearing reproductive organs, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Permanent sterilisation of the participant's sole partner (e.g. vasectomy) is also accepted.

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in those not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

***Complete abstinence (defined as refraining from heterosexual intercourse) must be in line with the preferred and usual lifestyle of the participant. Barrier contraception, periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation methods), withdrawal and progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action are not acceptable methods of contraception.

Exclusion Criteria:

* • Previous ischaemic heart disease (ST or non-ST myocardial infarction, Q3-risk >20, stable angina, unstable angina, stroke)

  * Any current or past history of malignancy, excluding squamous cell skin cancers
  * Concurrent opportunistic infection or other co-morbidity likely to occur during the trial e.g.

malabsorption syndromes, autoimmune disease

* Any contraindication to receipt of BHIVA recommended combination antiretrovirals
* Current treatment with injectable ART
* HTLV-1 co-infection
* Any evidence of major antiretroviral resistance mutations
* Evidence of HBV infection requiring treatment (HBsAg+, or HBcAb+ without HBsAb+)
* Evidence of HCV infection (HCVAg+ and/or HCV RNA detected)
* Individuals at high risk from severe Covid-19 disease who may be defined in accordance with NHSE guidance as vulnerable and shielded (as per the view of participant's physician)
* Current or planned systemic immunosuppressive therapy (inhaled and topical corticosteroids are allowed)
* Participation in another research study involving receipt of an investigational medicinal product (IMP) in the 3 months preceding enrolment or 5 half-lives of the investigational medicinal product, whichever is longer, or planned participation during the study period (concurrent observational studies are allowed)
* History of anaphylaxis or severe adverse reaction to antibody infusions, or hypersensitivity to GS-2872 or GS-5423 or to any constituent products or excipients thereof
* History of anaphylaxis or severe adverse reaction to any previous vaccine
* A history of thrombosis with thrombocytopaenia syndrome (TTS) following vaccination with any adenoviral vector vaccines
* A history of anti-phospholipid syndrome
* A history of heparin-induced thrombocytopenia
* A history of cerebral venous sinus thrombosis
* Any history of other bleeding or clotting disorders of clinical significance according to the investigator's discretion
* Known anti-PF4 antibody positivity
* Treatment with IV immunoglobulin or other monoclonal antibody treatments planned during the duration of the trial
* Clinically significant abnormal blood test results at screening including

  1. Moderate to severe hepatic impairment as defined by significant liver impairment with evidence of advanced fibrosis or cirrhosis with decompensation
  2. ALT >5 x ULN
  3. eGFR <601
  4. uPCR >30 mg/mmol
  5. INR >1.5
* Evidence of organ dysfunction or any clinically significant deviation from normal in medical history, physical examination and/or vital signs that the investigator believes is a preclusion from enrolment into the study
* Active alcohol or substance use that, in the investigator's opinion, will prevent adequate adherence with study requirements
* Insufficient venous access that will allow scheduled blood draws as per protocol
* Concern regarding likelihood of participant not taking precautions to prevent HIV transmission during treatment interruption period
* Pregnancy, lactation or intending to become pregnant
* Participants unable to be followed closely for geographic, social or psychological reasons
* Participants unable to adequately understand written or verbal English to appropriately consent to the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Fold change in T cell immune response to the HIV Gag protein | Baseline and 12 weeks after ATI
  The geometric mean of the fold-change (GMFC) will be compared between Arm C compared to Arm A; and Arm C compared to Arm B.

SECONDARY OUTCOMES:
Safety Assessment | From enrollment until 16 weeks after restarting ART after ATI
  Occurrence of Serious Adverse Events for the whole study duration.
Safety Assessment | From enrollment until 16 weeks after ART restart after ATI
  Number of participants with adverse events (not including SAEs)
HIV viral control | Weeks 12 and weeks 24 after ATI
  % of participants with undetectable plasma viral load
Immunological correlation of virological remission | Week 12 and week 24 after ATI
  CD4 T cell counts and CD8:CD4 ratios
Immunological correlates of virological remission | Weeks 12 and 24 after ATI
  HIV specific T cell immune response using multiple assays
BNAb plasma concentration | Weeks 12 and 24 after ATI
  bNAb maximum plasma concentration (Cmax)
ART plasma concentration | Week 12 and week 24 after ATI
  Maximum plasma concentration (Cmax) of ART
Vaccine specific response | Weeks 12 and 24 after ATI
  Proportion of participants that develop T cell response to HIVconsv immunogens
HIV reservoir assessment | Weeks 12 and 24 after ATI
  Measures of HIV reservoirs
bNAb escape | Weeks 12 and 24 after ATI
  Proportion of participants with bNAb resistance
T cell escape | Weeks 12 and 24 after ATI
  Proportion of participants with T cell escape mutations

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Guys and St Thomas' NHS Trust, London
  - St Mary's Clinical Trial Unit, London
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford

IPD SHARING:
Plan to Share IPD: No
The aim is to provide a summary of the results or a link to summary results within the trial registration record. Fully anonymised results will be published in peer reviewed papers and presented at conferences